CLINICAL TRIAL: NCT01585090
Title: Effect of Ankle Position and Pelvic Floor Muscle Force With Relaxation of Pelvic Floor Muscles Syndrome
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nahid golmakani, faculty member, Mashhad University of Medical Sciences
Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 89094
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Pelvic Floor Muscle Syndrome
Keywords: Ankle positions; pelvic floor muscles strength; relaxation of pelvic floor muscles syndrome; doing strengthening exercises of pelvic floor muscles

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- passive ankle dorsi ﬂexion (Experimental): doing strengthening exercises of PFM in standing position with passive ankle dorsi ﬂexion (on wooden surface with 15 degree angle)
  Interventions: Other: doing strengthening exercises of pelvic floor muscles
- active ankle plantar ﬂexion with arm up (Experimental): doing strengthening exercises of PFM in standing position with active ankle plantar ﬂexion with arm up (standing on toe)(n=20) and horizontal standing position
  Interventions: Other: doing strengthening exercises of pelvic floor muscles
- horizontal standing position (No Intervention): doing strengthening exercises of PFM in standing position with horizontal standing position
  Interventions: Other: doing strengthening exercises of pelvic floor muscles

INTERVENTIONS:
Other: doing strengthening exercises of pelvic floor muscles

SUMMARY:
Strengthening exercises of Pelvic Floor Muscles (PFM) is the first line treatment for female pelvic floor dysfunction. Actually the best position to facilitate PFM force is controversial in different studies. The aim of this study is to assess the effect of ankle positions on pelvic ﬂoor muscle force during PFM exercises.

This clinical trial study was carried out on 58 women aged 25-55 years with relaxation of pelvic floor muscles who referred to women's clinic of educational hospitals of Mashhad University of Medical Sciences in 1389. After clinical examination and confirmation of pelvic floor muscle relaxation, women were randomize divided into 3 groups, doing strengthening exercises of PFM in standing position with passive ankle dorsi ﬂexion (on wooden surface with 15 degree angle)(n=20), active ankle plantar ﬂexion with arm up (standing on toe)(n=20) and horizontal standing position (n=19) for 8 weeks. PFM exercises were instructed to women by using a pamphlet and face to face education. They were followed up every two week by telephone call and were asked to refer to women's clinic after 4 & 8 weeks. Pelvic floor muscles strength was assessed with brink score before and after intervention. Data analyzed by using analytic-descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* age 25-55
* bma 20-30
* women with relaxation of pelvic floor muscles syndrome in ph.ex and inspection

Exclusion Criteria:

* severe deformity in knee joint and ankle
* regular exercise or yoga
* severe or moderate vaginal atrophy

Ages: 25 Years to 55 Years | Sex: Female
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
pelvic floor muscles force